CLINICAL TRIAL: NCT00799591
Title: French Prospective Observational Study In Intensive Care Unit (ICU) Patients Treated With Tigecycline
Brief Title: French Study In ICU Patients Treated With Tigecycline
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 3074A1-4448; B1811030
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Results first posted 2011-12-19 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-09

CONDITIONS: Bacterial Infections
Keywords: Registre MONTRAVERS
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Intensive Care
  Interventions: Other: Observational study so no intervention in the patient.

INTERVENTIONS:
Other: Observational study so no intervention in the patient. — Observational study so no intervention in the patient.

SUMMARY:
This study will describe clinical outcome and safety data collected prospectively in subjects hospitalized in an intensive care unit (ICU) presenting with an infection for which treatment with tigecycline, alone or in combination, is planned. Data will be collected only from subjects providing informed consent.

DETAILED DESCRIPTION:
Healthcare visit.

Extension Rationale:

In order to perform the necessary corrective actions required and to secure database consistency, we request an extension for posting of Basic Results due 26-May-2011 for protocol 3074A1-4448 (B1811030), NCT00799591. Our proposed submission date is 14-Sept-2011.

Pfizer acquired Wyeth on October 16, 2009. With regard to this study, our reconciliation of data identified some discrepancies in data listed in the Project database (managed by the CRO) and the Safety Database (managed by Pfizer). We are taking corrective action which involves: sending queries to investigators, collecting corrective signed forms, and implementing changes within the database. We are requesting this extension to complete that work so that the data can be treated as final and the CSR can be completed.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women (18 years).
* Subjects hospitalized in a medical or surgical intensive care unit (ICU) (on the day of enrolment in the study).
* Subjects treated with tigecycline (first, second or third line), said treatment freely chosen by the participating physician, prior to enrollment in the study.

Exclusion Criteria:

* Subjects participating in another biomedical research study.
* Patient (or legal representative) who has not dated or signed informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Paris, France

REFERENCES:
- [Derived] Bassetti M, Eckmann C, Bodmann KF, Dupont H, Heizmann WR, Montravers P, Guirao X, Capparella MR, Simoneau D, Sanchez Garcia M. Prescription behaviours for tigecycline in real-life clinical practice from five European observational studies. J Antimicrob Chemother. 2013 Jul;68 Suppl 2:ii5-14. doi: 10.1093/jac/dkt140. PMID 23772047
- [Derived] Guirao X, Sanchez Garcia M, Bassetti M, Bodmann KF, Dupont H, Montravers P, Heizmann WR, Capparella MR, Simoneau D, Eckmann C. Safety and tolerability of tigecycline for the treatment of complicated skin and soft-tissue and intra-abdominal infections: an analysis based on five European observational studies. J Antimicrob Chemother. 2013 Jul;68 Suppl 2:ii37-44. doi: 10.1093/jac/dkt143. PMID 23772045
- [Derived] Montravers P, Bassetti M, Dupont H, Eckmann C, Heizmann WR, Guirao X, Garcia MS, Capparella MR, Simoneau D, Bodmann KF. Efficacy of tigecycline for the treatment of complicated skin and soft-tissue infections in real-life clinical practice from five European observational studies. J Antimicrob Chemother. 2013 Jul;68 Suppl 2:ii15-24. doi: 10.1093/jac/dkt141. PMID 23772042
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3074A1-4448&StudyName=French%20Study%20In%20ICU%20Patients%20Treated%20With%20Tigecycline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective observational study, non-comparative, conducted in 26 French Intensive Care Units (ICUs). Patients who were hospitalized in ICUs and presented with complicated infections of skin or soft tissues or complicated intra-abdominal infections and who met the inclusion criteria of the study were included in the study.
Groups:
- Tigecycline: Use and dosage recommendations for tigecycline (Tygacil®) were on the basis of the approved Summary of Product Characteristics (SmPC) and adjusted solely according to medical and therapeutic necessity. Tigecycline powder for solution for intravenous (IV) infusion could be administered with an initial loading dose of 100 milligrams (mg) followed by 50 mg administered IV (over 30 to 60 minutes) every 12 hours for 5 to 14 days.
Period: Overall Study
Arm/Group | Tigecycline
Started | 156
Completed | 90
Not Completed | 66
Not completed — De-escalation of doses | 20
Not completed — Death | 14
Not completed — Technical failure | 12
Not completed — Resistant germ | 11
Not completed — New infection | 4
Not completed — Resistance germ and technical failure | 2
Not completed — Persistance of fever undetermined origin | 1
Not completed — Antibiotic changed, no apparent reason | 1
Not completed — Infectious origin not probable | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tigecycline
Number analyzed (Participants) | 156
Age Continuous [Mean (Standard Deviation); unit: years] | 60.1 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 100
Percentage of participants per type of infection: Intra-abdominal [Number; unit: percentage of participants] — Nosocomial=hospital acquired infection. Participants may be represented in > 1 category. Infection N=88, Peritonitis N=68, Localization N=88.
  percentage of participants
    Infection: Nosocomial | 69.3
    Infection: Community | 30.7
    Peritonitis: Generalized | 63.2
    Peritonitis: Abscess without peritonitis | 22.1
    Peritonitis: Localized | 14.7
    Localization ≥ 10%: Colon | 37.5
    Localization ≥ 10%: Other | 12.5
Percentage of participants per type of infection: Infection of skin and soft tissue [Number; unit: percentage of participants] — Nosocomial=hospital acquired infection. Participants may be represented in > 1 category. Infection N=29, Dermo-panniculis N=29, Localization N=17.
  percentage of participants
    Infection: Nosocomial | 69.0
    Infection: Community | 31.0
    Dermo-panniculis | 96.6
    Localization ≥ 10%: Abdomen | 52.9
    Localization ≥ 10%: Head and neck | 29.4
    Localization ≥ 10%: Perineum | 11.8
Percentage of participants per type of infection: Other infections [Number; unit: percentage of participants] — Nosocomial=hospital acquired infection. Participants may be represented in > 1 category. Infection N=56, Localization N=56.
  percentage of participants
    Infection: Nosocomial | 89.3
    Infections: Community | 10.7
    Localization ≥ 10%: Lung | 67.9
    Localization ≥ 10%: Miscellaneous | 32.1
Mean Simplified Acute Physiology Score II (SAPSII): Integer score [Mean (Standard Deviation); unit: scores on a scale] — Severity of disease measurement 24 hours after ICU admission based on 17 variables. Result values transformed to an integer point score from 0 (less severe disease state) to 163 (more severe disease state) and can also be used to calculate a corresponding mortality between 0% (no predicted mortality) and 100% (greatest predicted mortality). N=147
  scores on a scale | 43.3 (16.4)
Mean Sepsis-related Organ Failure Assessment (SOFA) score [Mean (Standard Deviation); unit: scores on a scale] — Assess extent of organ function or rate of failure during ICU admission. Based on scores for 6 systems (respiratory, cardiovascular, hepatic, coagulation, renal, and neurological) graded from 0 (normal) to 4 (most abnormal) with a potential total score of 0 to 24; higher score indicates greater system abnormality.
  scores on a scale | 7.0 (4.5)
Percentage of participants per reason for choice of treatment with Tigecycline [Number; unit: percentage of participants] — Participants may be represented in > 1 category. Multi-resistant bacteria (MRB).
  percentage of participants
    Polymicrobial infection | 55.1
    MRB suspected or identified | 40.4
    Renal impairment | 17.9
    Multiple sites | 15.4
    Failure of previous treatment | 12.2
    Allergy or intolerance to other antiobiotics | 9.6
    Rescue medication | 8.3
    Other | 6.4
Percentage of participants per co-morbid (concomitant) diseases [Number; unit: percentage of participants] — Participants may be represented in > 1 category. Immunosuppression (Immuno).
  percentage of participants
    Diabetes mellitus | 5.1
    Non-insulin dependent diabetes | 14.1
    Chronic renal failure | 10.3
    Chronic hepatic failure Type A | 80.0
    Chronic hepatic failure Type C | 20.0
    Immuno > 10%: Cancer | 53.8
    Immuno > 10%: Use of corticoids | 15.4
    Immuno > 10%: Corticoids plus other Immuno | 15.4
    Immuno > 10%: Other Immuno | 13.5
Percentage of participants with antibiotic treatment(s) taken 30 days prior to Tigecycline treatment [Number; unit: percentage of participants]
  Treatment within 30 days prior=No | 7.1
  Treatment within 30 days prior=Yes | 92.9
Percentage of participants with microbiological sampling results: positive blood culture [Number; unit: percentage of participants] — Microbiological sampling results categorized as a positive blood culture (presence of infection); N=145
  percentage of participants | 11.7
Percentage of participants with microbiological sampling results: direct examination [Number; unit: percentage of participants] — Microbiological sampling results categorized according to direct examination (identification of the class of germs). Participants may be represented in >1 category. N=87
  percentage of participants
    Gram negative bacilli | 59.8
    Gram positive cocci | 47.1
    Polymicrobial | 33.3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Per Clinical Outcome (Success, Failure, or Undetermined) at End of Treatment (EOT)
Description: Clinical Success: lack of need to use new antibiotic or a surgical treatment not initially planned for initial infection. Failure: persistence of initial infection (required change of antibiotic or surgery), death related to infection (>48 hours after start of treatment with tigecycline), or premature cessation of treatment due to treatment-related Adverse Event. Undetermined: insufficient data for assessment, death not directly related to initial infection, death within first 48 hours of start of treatment with tigecycline, or additional antibiotic treatment for other than initial infection.
Time Frame: End of Treatment (on the day of last dose of study treatment) or up to 25 months
Population: Intent-to-Treat (ITT): all participants included in the study who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tigecycline
Number analyzed (Participants) | 156
percentage of participants
  Success | 59.6 [51.5 to 67.4]
  Clinical Failure - deaths | 2.6 [0.7 to 6.4]
  Clinical Failure - other criteria | 15.4 [10.1 to 22.0]
  Undetermined | 22.4 [16.2 to 29.8]

2. Primary Outcome: Percentage of Participants Per Clinical Outcome (Success, Failure, or Undetermined) at Follow-up Visit
Description: as for outcome 1
Time Frame: Follow-up Visit (7 days after last dose or at hospital discharge whichever occurred within 7 days after last dose) or up to 25 months
Population: ITT population; N=number of participants with analyzable data at observation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tigecycline
Number analyzed (Participants) | 145
percentage of participants
  Success | 53.1 [44.6 to 61.4]
  Clinical Failure | 22.1 [15.6 to 29.7]
  Undetermined | 24.8 [18.0 to 32.7]

3. Secondary Outcome: Percentage of Participants Per Tigecycline Loading Dose and Maintenance Dose
Description: Tigecycline powder for solution 50 milligrams (mg) for intravenous (IV) infusion could be administered with an initial loading dose of 100 mg followed by 50 mg administered IV (over 30 to 60 minutes) every 12 hours for 5 to 14 days. Use and dosage recommendations for tigecycline (Tygacil®) were on the basis of the approved Summary of Product Characteristics (SmPC) and adjusted solely according to medical and therapeutic necessity.
Time Frame: Baseline (Inclusion) through last dose of study treatment or up to 25 months
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Tigecycline
Number analyzed (Participants) | 156
percentage of participants
  Loading dose: 100 mg | 97.4
  Loading dose: Other | 2.6
  Maintenance dose: 50 mg twice a day | 93.6
  Maintenance dose: 50 mg twice a day + Other | 0.6

4. Secondary Outcome: Mean Duration (Days) of Treatment With Tigecycline
Time Frame: Baseline (Inclusion) through last dose of study treatment or up to 25 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tigecycline
Number analyzed (Participants) | 156
days | 10.2 (8.8)

5. Secondary Outcome: Percentage of Participants (> 10%) With Use of Other Antibiotics in Combination With Tigecycline Who Had Clinical Success at EOT
Description: Combinations of antibiotic treatments for participants treated with clinical success with tigecycline. Clinical success defined as lack of need to use new antibiotic or a surgical treatment not initially planned for initial infection.
Time Frame: Baseline (Inclusion), End of Treatment (on the day of last dose of study treatment) or up to 25 months
Population: ITT population; N=number of participants treated with combinations of antibiotics with analyzable data at observation.
Measure: Number; unit: percentage of participants
Arm/Group | Tigecycline
Number analyzed (Participants) | 93
percentage of participants
  Aminoglycosides | 22.6
  Aminoglycosides: Amikacin | 14.0
  Penicillins | 15.1
  Penicillins: Piperacillin / Tazobactam | 9.7

6. Secondary Outcome: Percentage of Participants (> 10%) With Use of Other Antibiotics in Combination With Tigecycline Who Had Clinical Success at Follow-up Visit
Description: as for outcome 5
Time Frame: Baseline (Inclusion), Follow-up Visit (7 days after last dose or at hospital discharge whichever occurred within 7 days after last dose) or up to 25 months
Population: ITT population; N=number of participants treated with combinations of antibiotics with analyzable data at observation.
Measure: Number; unit: percentage of participants
Arm/Group | Tigecycline
Number analyzed (Participants) | 77
percentage of participants
  Aminoglycosides | 23.4
  Aminoglycosides: Amikacin | 14.3
  Penicillins | 15.6
  Penicillins: Piperacillin / Tazobactam | 10.4

7. Secondary Outcome: Percentage of Participants With Microbiological Sampling Results During Treatment Phase With Tigecycline: Positive Blood Culture
Description: Microbiological sampling results categorized as a positive blood culture (presence of infection).
Time Frame: Post-baseline (Day 1) through last dose of study treatment or up to 25 months
Population: ITT population. N=number of participants with analyzable data at observation.
Measure: Number; unit: percentage of participants
Arm/Group | Tigecycline
Number analyzed (Participants) | 148
percentage of participants | 8.8

8. Secondary Outcome: Percentage of Participants With Microbiological Sampling Results During Treatment Phase With Tigecycline: Direct Examination
Description: Microbiological sampling results categorized according to direct examination (identification of the class of germs).
Time Frame: Post-baseline (Day 1) through last dose of study treatment or up to 25 months
Population: ITT population. N=number of participants with analyzable data at observation; participants may be represented in >1 category.
Measure: Number; unit: percentage of participants
Arm/Group | Tigecycline
Number analyzed (Participants) | 33
percentage of participants
  Gram negative bacilli | 66.7
  Gram positive cocci | 27.3
  Polymicrobial | 18.2
  Gram positive bacilli | 3.0

ADVERSE EVENTS:
Time Frame: Baseline (Inclusion) through 7 days after end of study treatment or up to 25 months
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tigecycline
Serious Adverse Events (participants affected / at risk) | 26/156
Other Adverse Events (participants affected / at risk) | 9/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tigecycline (N=156)
Multiorgan failure (General disorders) | 9
Drug resistance (General disorders) | 1
Amount of liquid intra-abdominal localized (Gastrointestinal disorders) | 2
Colitis ischaemia (Gastrointestinal disorders) | 1
Intestinal infarction (Gastrointestinal disorders) | 1
Pancreatic necrosis (Gastrointestinal disorders) | 1
Small intestine obstruction (Gastrointestinal disorders) | 1
Septic shock (Infections and infestations) | 6
Purulent discharge (Infections and infestations) | 1
Haemorrhage (Vascular disorders) | 1
Atrio ventricular dissociation (Cardiac disorders) | 1
Carotid artery dissection (Nervous system disorders) | 1
Hallucination (Psychiatric disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Lack of efficacy of the drug (ineffectiveness of the drug) (General disorders) | 1
Hemorrhagic shock (Shock due to an haemorrhage) (Vascular disorders) | 1
Arterial injury (lesion of an artery) (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tigecycline (N=156)
Vomiting / Nausea (Gastrointestinal disorders) | 3
Fungal infection (Infections and infestations) | 2
Cholestasis (Hepatobiliary disorders) | 3
Renal failure acute (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.